CLINICAL TRIAL: NCT01838161
Title: Project INSPIRE: Improving Adolescent Vaccination in Appalachian Kentucky
Brief Title: Improving Adolescent Vaccination in Appalachian Kentucky
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-0026-P4S
Record Dates: First submitted 2013-04-04; First posted 2013-04-23 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Adolescent Immunization
Keywords: adolescents; immunizations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part I (Active Comparator): Interview questions will focus on reticence to vaccinate children.
  Interventions: Behavioral: Part I
- Part II (Experimental): We will pilot the vaccination vignettes in a health department (clinical) setting with eligible parents of adolescents.
  * a pretest survey
  * the video vignette
  * and a post-test survey measuring intention to receive appropriate adolescent vaccines
  Interventions: Behavioral: Part II
- Part III (Experimental): * enhanced video educational intervention (video vignettes + standard of care vaccine event)
  * standard of care vaccination event
  Interventions: Behavioral: Part III

INTERVENTIONS:
Behavioral: Part II — Parents will be exposed to an educational video intervention if they are enrolled in this intervention condition.
  Arms: Part II
Behavioral: Part III — •video educational
  Other Names: Video Education
  Arms: Part III
Behavioral: Part I — Parental Interviews
  Arms: Part I

SUMMARY:
The proposed project develops a community and school-based intervention to enhance understanding of the importance all age-appropriate vaccinations, and uses an innovative, comprehensive approach (Project INSPIRE - Instilling Necessary Sickness Prevention with Immunizations Reaching Everyone) to ensure that all parents of adolescents are advised of all age-appropriate vaccines for sickness prevention. The investigator will develop a novel set of targeted video vignette persuasive informational decision aids (including target population representatives) to enhance lay understanding of recommended adolescent (or catch-up) vaccines. The Investigator will also partner with school districts to develop a replicable social marketing vaccination event program (Project INSPIRE) to encourage parents and teens to publicly vaccinate at community events and during drop-in school nursing clinic hours. The project will test the efficacy of the video-based health education intervention + standard of care to ideal standard of care (social marketing vaccination event program) approaches to immunize adolescents in this region.

DETAILED DESCRIPTION:
This is not an interventional study in which subject will be given a investigator drug or device.

Part I of the INSPIRE intervention development will involve formative research interviews conducted with parents of adolescents. Interview questions will focus on reticence to vaccinate children. Participants will be a convenience sample recruited through contacts in local public health departments and community nurses recruited by flyer and the research study coordinators (UK study personnel). Interview sessions will be scheduled in advance and will take approximately 30 minutes.

Part II of the INSPIRE intervention development will be evaluated in a small clinic-based pilot study using the same pre-test/post-test intervention design as in the planned (Part III) trial. For the pilot testing, the investigators will pilot the vaccination vignettes in a health department (clinical) setting with eligible parents of adolescents. Eligible parents who are coming in for non-acute care appointments will be asked by a research nurse to enroll in a research study. The Investigator will then administer a pretest survey, expose participants (parents) to vignette condition using the iPad in the clinic, and a post-test survey measuring intention to receive appropriate adolescent vaccines for their child as well as perceived message effectiveness (for the vignette). At the conclusion of the study, the research personnel administering the study will refer the adolescent to the clinic staff who will offer adolescent vaccines at the conclusion of the study (and/or a cue to schedule an appointment for the adolescent to visit the clinic) and will be able to examine actual behavior by receiving informed consent (from parents and adolescent) for limited medical record review (to track adolescent receipt of vaccinations). The Investigator will perform this pilot study in one Kentucky River Area District health department clinic with 30 parents. This method has been used to pilot past interventions, and it is expected that this allow us to correct for any problems in either the design of the survey assessment or the intervention. If needed, the investigator can tweak the intervention and re-pilot using the same procedures before the randomized controlled trial. This pilot test will also provide the advantage of assuring us that the intervention procedure can translate to the clinic setting. The Investigator has experience with this translation from our 1-2-3 Pap video intervention which the investigators began in social settings (recruiting people at school and other community events) and moved into the clinic setting for dissemination.

Part III of the INSPIRE project will be evaluated in a site-based group randomized controlled trial design, with individual-level randomization also occurring within the intervention group. Community vaccination clinic and health education sites (staffed by local health department contracted personnel and project nurses) in the intervention and control conditions will be matched on percentage of free/reduced school lunch and relevant demographics. At the end of Year 1, one health site in each pair will be randomized to the enhanced video educational intervention (video vignettes + standard of care social marketing vaccine event) or a standard of care vaccination campaign (standard of care health department vaccine event) comparison group. Individuals in the intervention group randomized condition also will be randomized when recruitment occurs in non-school based locations. Assessments will be conducted using Automated iPad Audio Assisted Interviewing techniques at pretest, immediate post-test, and then medical record review at 1 month and 9 month follow-up points. The medical record review will entail examining the medical record for each adolescent vaccine received by the patient. Thus, the investigators will be able to examine behavior change (i.e., receipt of vaccination) for each of the different vaccine types and their single or multi-dose outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians with legal custody of a minor child
* Parents of children 11-18 years of age.

Exclusion Criteria:

* Parents under the age of 18
* Allergy to vaccinations
* Parent has made an informed decision not to vaccinate their child

Ages: 11 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Part I - Parent Interviews | 1 year
  Interview questions will focus on reticence to vaccinate children. Participants will be a convenience sample recruited through contacts in local public health departments, community nurses and the research study coordinators.

SECONDARY OUTCOMES:
Part II - Intention to Vaccinate | 1 Year
  The investigator will pilot the vaccination vignettes in a health department (clinical) setting with eligible parents of adolescents. The Investigator will then expose parents to vignette condition using the iPad, administer a pretest survey, the video vignette, and a post-test survey measuring intention to receive appropriate adolescent vaccines for their child as well as perceived message effectiveness (for the vignette).

OTHER OUTCOMES:
Part III - Site-based group randomized controlled trial design - Vaccination outcomes | 1 year
  Community vaccination clinic sites in the intervention and control conditions will be matched on percentage of free/reduced school lunch and relevant demographics. Randomization will occur at the group and individual level. One site in each pair will be randomized to the enhanced video educational intervention condition (within this group individuals will be randomized to video vignettes + standard of care vaccine education or the standard of care vaccine education) or a standard of care (standard of care vaccine education) comparison group. The medical record review will allow us to examine behavior change (i.e., receipt of age-appropriate vaccinations) for each of the different vaccine types and their single or multi-dose outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Elisia Cohen, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen, E. L. and K. J. Head (2014).